CLINICAL TRIAL: NCT06146972
Title: Efficacy Study of Iguratimod Combined With Tofacitab in Patients With RF Positive/Negative Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yanfeng Hou (Other)
Responsible Party: Sponsor-Investigator, Yanfeng Hou, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZPK2021Z0629
Record Dates: First submitted 2023-08-09; First posted 2023-11-27 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Rheumatoid Arthritis; Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod; tofacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RF positive group (Experimental): Iguratimod (25mg per tablet) 25mg twice daily plus tofacitinib (5mg per tablet) 5mg twice daily for 24 weeks.
  Interventions: Drug: Iguratimod
- RF negative group (Experimental): Iguratimod (25mg per tablet) 25mg twice daily plus tofacitinib (5mg per tablet) 5mg twice daily for 24 weeks.
  Interventions: Drug: Iguratimod

INTERVENTIONS:
Drug: Iguratimod — Iguratimod 25mg bid + tofacitinib 5mg bid
  Other Names: tofacitinib

SUMMARY:
Rheumatoid arthritis (RA) is a chronic progressive autoimmune disease with predominantly joint involvement. To compare the efficacy and difference between elamod and tofacitib in the treatment of rheumatoid factor-positive and negative rheumatoid arthritis in RA patients with poor outcome after csDMARDs dosing, in order to better inform the clinical management.

DETAILED DESCRIPTION:
This is an open, controlled, interventional clinical study enrolling patients with active RA who meet the following entry row criteria, and treating patients with IGU 25 mg bid + tofacitinib 5 mg bid for the intervention. The screening period was defined as the screening visit was conducted within 1 month prior to the baseline visit, and efficacy and safety assessments were performed at time points 0, 4, 12, 18, and 24 weeks from the time the subject was treated with the study protocol (see efficacy and safety endpoints for details), and study subjects were asked to come to the hospital for follow-up within ±3 days of the corresponding follow-up point.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-65 years old
2. Body weight not less than 40kg
3. Patients with a clear diagnosis of rheumatoid arthritis (RA) who meet the diagnostic criteria for RA introduced by the ACR in 1987 or ACR\EULAR in 2010
4. Joint function grade II-III
5. Active rheumatoid arthritis (defined as active rheumatoid arthritis if the following three conditions are met: ① ≥ 6 joints swollen [66 joints count]

   ② ≥ 6 joints tenderness [68 joints count]

   ③Erythrocyte sedimentation rate (ESR) > 28 mm/h or C-reactive protein (CRP) > 1.0 mg/dL)
6. The Patients have been treated with csDMARDs for ≥ 3 months and have been treated with stable doses of csDMARDs for 4 consecutive weeks prior to study entry, with poor therapeutic outcomes and are being considered for treatment with a combination of biologics (bDMARDs) (according to the 2018 China Rheumatoid Arthritis Treatment Guidelines, poor outcomes, i.e., no significant improvement in RA disease activity within 3 months or failure to achieve treatment goals within 6 months)
7. Subjects must be able and willing to perform subcutaneous (SC) injections on their own, or a qualified person must be available to perform SC injections
8. If taking glucocorticosteroids, prednisone should be ≤10mg or other hormone at a dose equivalent to prednisone and the dose should be kept constant for at least 28d
9. Understand the purpose of the trial and the test procedures and sign a written informed consent form voluntarily

Exclusion Criteria:

1. Patients who have used potent immunosuppressants (such as cyclophosphamide, cyclosporine, azathioprine, etc.), tripterygiam glycosides and so on that affect the evaluation of efficacy in previous rheumatoid arthritis treatment , and who have stopped taking them for less than 4 weeks
2. History of allergy to relevant test drugs
3. Previously treated with bDMARDs
4. Subject has recently received a live vaccine, or plans to use any live vaccine during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-24 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
ACR20 | 24 weeks
  ACR20 is the gold standard for the degree of disease remission in RA. The specifics are: according to the ACR criteria, the patient's joint tenderness count (TJC) and joint swelling count (SJC) improved by ≥20%, and at least three of the following five parameters improved by ≥20%:① Pain Visual Analog Scale (VAS) ② the Patient Global Assessment (PGA) ③ Physician Global Assessment (MDGA) ④ Health Assessment Questionnaire disability index (HAQ DI) score ⑤ Acute-phase reactants (ESR or CRP).
ACR50 | 24 weeks
  The specifics are: according to the ACR criteria, the patient's joint tenderness count (TJC) and joint swelling count (SJC) improved by ≥50%, and at least three of the following five parameters improved by ≥50%:① Pain Visual Analog Scale (VAS) ② the Patient Global Assessment (PGA) ③ Physician Global Assessment (MDGA) ④ Health Assessment Questionnaire disability index (HAQ DI) score ⑤ Acute-phase reactants (ESR or CRP).
DAS28 (ESR) | 24 weeks
  Disease activity was assessed by calculating the DAS28 score; ≤2.6 was considered remission, >2.6 and ≤3.2 was considered low disease activity, >3.2 and ≤5.1 was considered moderate disease activity, and >5.1 was considered high disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Yanfeng Hou, Dr., Study Director — Yanfeng Hou
Locations (1):
- Yanfeng Hou, Jinan, Shandong, China